CLINICAL TRIAL: NCT06194929
Title: Phase 1b/2 Trial of Defactinib and Avutometinib, With or Without Encorafenib, for the Treatment of Patients With Brain Metastases From Cutaneous Melanoma
Brief Title: Defactinib and Avutometinib, With or Without Encorafenib, for the Treatment of Patients With Brain Metastases From Cutaneous Melanoma
Acronym: DETERMINE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI168254
Record Dates: First submitted 2023-12-20; First posted 2024-01-08 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Cutaneous Melanoma; Brain Metastases
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — defactinib; encorafenib

STUDY DESIGN:
Intervention Model Description: Cohort A will evaluate the hypothesis that avutometinib and defactinib will have clinical benefit in terms of response rate and/or for prolonging organ specific PFS in patients with cutaneous melanoma and at least one untreated brain metastases after at least one line of immunotherapy (Cohort A), compared to historical controls.
  Cohort B will evaluate the hypotheses that avutometinib, defactinib, and encorafenib will have clinical benefit in terms of response rate and/or for prolonging organ specific PFS in patients who have received at least one prior line of immunotherapy and also may have received at least one line of prior BRAF/MEK therapy, compared to historical controls. Cohort B will also include a limited dose escalation cohort using a BOIN design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase II, Defactinib and Avutometinib (Cohort A) (Experimental): Avutometinib will be administered at 3.2 mg biweekly orally (e.g., Monday/Thursday, Tuesday/Friday, or Wednesday/Saturday) for 3 weeks, followed by a 1-week rest period, in each 4-week (28-day) cycle.
  Defactinib will be administered at 200 mg twice a day orally for 3 weeks, followed by a 1-week rest period, in each 4-week (28-day) cycle.
  Interventions: Drug: Defactinib; Drug: Avutometinib
- Phase Ib, Defactinib, Avutometinib, and Encorafenib (Cohort B) (Experimental): Avutometinib will be administered at 3.2 mg biweekly orally (e.g., Monday/Thursday, Tuesday/Friday, or Wednesday/Saturday) for 3 weeks, followed by a 1-week rest period, in each 4-week (28-day) cycle.
  Defactinib will be administered at 200 mg twice a day orally for 3 weeks, followed by a 1-week rest period, in each 4-week (28-day) cycle.
  Encorafenib will be administered orally to a small cohort to a limited dose finding cohort using a Bayesian optimal interval (BOIN) design to evaluate safety, toxicity, and recommended phase II dose for dosage of encorafenib when combined with avutometinib and defactinib.
  Dose escalation/de-escalation levels for Encorafenib:
  Dose Level -1: 225 mg Daily (three 75mg capsules) Dose Level 0: 300 mg Daily (four 75mg capsules) Dose Level 1: 450 mg Daily (six 75mg capsules)
  Interventions: Drug: Defactinib; Drug: Avutometinib; Drug: Encorafenib
- Phase II, Defactinib, Avutometinib, and Encorafenib (Cohort B) (Experimental): Avutometinib will be administered at 3.2 mg biweekly orally (e.g., Monday/Thursday, Tuesday/Friday, or Wednesday/Saturday) for 3 weeks, followed by a 1-week rest period, in each 4-week (28-day) cycle.
  Defactinib will be administered at 200 mg twice a day orally for 3 weeks, followed by a 1-week rest period, in each 4-week (28-day) cycle.
  Encorafinib will be administered orally at doses defined in the dose finding portion (225mg - 450mg) Daily continuously (days 1-28 of a 28 day cycle) for Cohort B.
  Interventions: Drug: Defactinib; Drug: Avutometinib; Drug: Encorafenib

INTERVENTIONS:
Drug: Defactinib — Defactinib will be administered at 200 mg twice daily orally per arm description.
Drug: Avutometinib — Avutometinib will be administered at 3.2 mg twice a week orally per arm description.
Drug: Encorafenib — Encorafinib administered orally per arm description.
  Arms: Phase II, Defactinib, Avutometinib, and Encorafenib (Cohort B); Phase Ib, Defactinib, Avutometinib, and Encorafenib (Cohort B)

SUMMARY:
The goal of this interventional clinical trial is to provide proof-of-principle data for the biologic activity of defactinib in combination with avutometinib in brain metastases from melanoma, and to define the potential role of the combination with mutant BRAF inhibitors or after BRAF/MEK inhibitors in BRAF V600E/K mutant tumors, in individuals with advanced melanoma who experience the development or progression of brain metastases after treatment with immune checkpoint inhibitors.

The main questions it aims to answer are:

* What is the preliminary response rate of defactinib and avutometinib in patients with RAS mutant, BRAF mutant, NF1 mutant, triple RAS/BRAF/NF1 wild type (wt) melanoma (including RAF fusions)?
* What is the safety and tolerability of the combination of defactinib, avutometinib, and encorafenib in patients with BRAF V600E/K mutant melanoma with at least one untreated brain metastases?
* What is the preliminary response rate of the three drug combination of defactinib, avutometinib, and encorafenib in patients with BRAF V600E/K mutant melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of informed consent.
* Provide written informed consent and comply with the study protocol as judged by the Investigator. Of note, If the subject has an impairment that prevents him/her from providing written consent, the site may follow local institutional procedures for obtaining consent.
* Histologically confirmed diagnosis of cutaneous melanoma with radiographically confirmed metastases to the brain.
* Must have a tumor with a known RAS, BRAF, or NF1 mutation or triple wildtype status using validated testing methods prior to enrollment. Cohorts will be assigned as follows:

  * Cohort A: RAS, BRAF, NF1, or triple wildtype
  * Cohort B: BRAF V600E or BRAF V600K
* Must have at least 1 untreated (no prior resection or radiation of the target lesion) parenchymal brain metastasis with minimal dimensions of ≥ 0.5 cm diameter and maximal dimensions ≤ 4 cm diameter, measured from a gadolinium enhanced MRI T1 sequence.

  * Note: Subject may have received prior resection or radiation therapy for prior brain metastases.
* Must have received at least 1 line of prior systemic immunotherapy.
* For Cohort B, may have received 1 or more lines of prior BRAF or MEK inhibitor therapy.
* An ECOG Performance Status of 0 or 1, or Karnofsky score >= 70
* Adequate bone marrow, organ function and laboratory parameters:

  * ANC ≥ 1.5 × 109/L;
  * Hemoglobin ≥ 9 g/dL with or without transfusions;
  * Platelets ≥100,000/mm2;
  * AST and ALT ≤ 2.5 × ULN; in patients with liver metastases ≤ 5 × ULN;
  * Total bilirubin ≤ 1.5 × ULN; NOTE: Patients with documented Gilbert syndrome or hyperbilirubinemia due to non-hepatic cause (e.g., hemolysis, hematoma) may be enrolled
  * Serum creatinine ≤ 1.5 × ULN; OR calculated creatinine clearance > 50 mL/min by Cockcroft-Gault formula; OR estimated glomerular filtration rate > 50 mL/min/1.73m2.
  * International normalized ratio (INR), prothrombin time (PT), or activated partial thromboplastin time (aPTT) as follows:

    * In the absence of therapeutic intent to anticoagulate the patient:

      * INR < 1.5 × ULN.
      * PT < 1.5 × ULN.
      * aPTT < 1.5 × ULN.
      * Adequate cardiac function with left ventricular ejection fraction ≥ 55% by echocardiography (ECHO) or multiple-gated acquisition (MUGA) scan.
* For women (any individual assigned female at birth) who are not postmenopausal (ie, < 2 years after last menstruation) or surgically sterile (absence of ovaries and/or uterus) and who are sexually active, must have a negative serum pregnancy test and agree to use a highly effective method of contraception for the duration of the study and for 90 days following the last dose of study drug.
* Male patients (any individual assigned male at birth) of reproductive potential must avoid pregnancy in partners who are women of childbearing potential, and such partners should not consider getting pregnant during the study and for at least 90 days after treatment is discontinued or longer if requested by local authorities. Male patients are considered to be of reproductive potential unless permanently sterile by bilateral orchidectomy or vasectomized with appropriate post-vasectomy documentation of absence of sperm in ejaculate.
* Adequate recovery to baseline or ≤ Grade 1 CTCAE v5 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy per the treating investigator. Exceptions include alopecia and peripheral neuropathy grade ≤ 2.

Exclusion Criteria:

* Receiving other investigational agents.
* Prior systemic anti-cancer therapy or any investigational therapy ≤ 28 days or within five half-lives prior to starting study treatment, whichever is shorter.
* Patients with symptomatic brain metastasis, defined as neurologic symptoms with localization attributable to an untreated brain metastases with severity >= Grade 2 by CTCAE criteria.
* History of allergy or hypersensitivity to any of the study treatments or any of their excipients.
* Inability to swallow and retain study treatment.
* Uveal or mucosal melanoma.
* History of or current leptomeningeal metastases.
* QTcF > 450 msec if male and QTcF > 470 msec if female.
* Any hemorrhage or bleeding event that is ≥ Grade 3 based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event (CTCAE) or Grade 2 intracranial hemorrhage within 4 weeks prior to the start of study treatment.
* Uncontrolled or severe cardiac disease (eg, history of unstable angina, myocardial infarction, coronary stenting, or bypass surgery within the last 6 months prior to initiation of study treatment), symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia (including atrial flutter/fibrillation), requirement for inotropic support or use of devices for cardiac conditions (eg, pacemakers/defibrillators), or hypertension (patients with systolic blood pressure [BP] of > 160 mm Hg or diastolic BP of > 100 mm Hg despite optimal medical management are to be excluded).
* History of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis, or symptomatic pleural effusion.
* Active, known, or suspected uncontrolled autoimmune disease, which required therapy in the past 2 years, including but not limited to systemic lupus erythematosus, Hashimotos thyroiditis, scleroderma, polyarteritis nodosa, or autoimmune hepatitis.
* Known HIV infection with a detectable viral load within 6 months of the anticipated start of treatment. Note: Participants on effective antiretroviral therapy with an undetectable viral load within 6 months of the anticipated start of treatment are eligible for this trial.
* Systemic active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination, radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), or hepatitis C. Note: Participants with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Participants positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* History of bleeding diathesis (irrespective of severity) in the absence of therapeutic anticoagulation.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection.
* Any condition that could make the patient noncompliant with the study procedures and/or study requirements, as judged by the Investigator.
* Active skin disorder that has required systemic therapy within the past 1 year.
* History of rhabdomyolysis.
* Concurrent ocular disorders:

  * Patients with history of glaucoma, history of retinal vein occlusion (RVO), predisposing factors for RVO, including uncontrolled hypertension, uncontrolled diabetes.
  * Patients with history of retinal pathology or evidence of visible retinal pathology that is considered a risk factor for RVO, intraocular pressure > 21 mm Hg as measured by tonometry, or other significant ocular pathology, such as anatomical abnormalities that increase the risk for RVO.
  * Patients with active or chronic, visually significant corneal disorders, other active ocular conditions requiring ongoing therapy or clinically significant corneal disease that prevents adequate monitoring of drug-induced keratopathy. Examples of visually significant corneal disorders include corneal degeneration, active or recurrent keratitis, and other forms of serious ocular surface inflammatory conditions. Visually significant corneal disorders do NOT include dry eyes, blepharitis, and uncomplicated corneal erosions.
* Patients with a history of hypersensitivity to any of the active (avutometinib, defactinib, encorafenib) or inactive ingredients of the investigational products.
* Exposure to medications (with or without prescriptions), supplements, herbal remedies, or foods with potential for drug-drug interactions with study interventions within 14 days prior to the first dose of study intervention and during the course of therapy, including:

  * Strong CYP3A4 inhibitors or inducers, due to potential drug-drug interactions with both avutometinib and defactinib.
  * Strong CYP2C9 inhibitors or inducers, due to potential drug-drug interactions with defactinib.
  * Strong P-glycoprotein (P-gp) inhibitors or inducers, due to potential drug-drug interactions with both avutometinib and defactinib.
  * Strong breast cancer resistance protein (BCRP) inhibitors or inducers, due to potential drug-drug interactions with avutometinib.
* Concomitant treatment with warfarin. Patients who require anticoagulation but cannot discontinue warfarin must be excluded from the study.
* Participants taking other prohibited medications in protocol, including anticancer therapy or investigational agents and colony-stimulating factors (CSFs). A washout period of prohibited medications for a period of at least five half-lives or as clinically indicated should occur before the start of treatment.
* The diagnosis of another malignancy within ≤ 2 years before study enrollment, except for those considered to be adequately treated with no evidence of disease or symptoms and/or will not require therapy during the study duration (i.e., basal cell or squamous cell skin cancer, carcinoma in situ of the breast, bladder or of the cervix, or low-grade prostate cancer with Gleason Score ≤ 6)
* Any other condition that would, in the Investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures (e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, [subjects may not receive the drug through a feeding tube], social/ psychological issues, etc.)
* Medical, psychiatric, cognitive, or other conditions that may compromise the subject's ability to understand the subject information, give informed consent, comply with the study protocol or complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2028-01-15 (Estimated); Study Completion 2030-01-15 (Estimated)

PRIMARY OUTCOMES:
Response rate defined as Partial Response (PR) + Complete Response (CR) using Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria of all measurable target lesions present at the time of enrollment on trial. | 6 months
  For Cohort A, the primary objective will be to evaluate preliminary response rate of defactinib and avutometinib in patients with RAS mutant, BRAF mutant, NF1 mutant, and triple RAS/BRAF/NF1 wild type (wt) melanoma (includes RAF fusions). Measurable target lesions to be defined as all untreated and measurable (≥ 0.5 cm by 2 dimensional diameter measurements) present at the time of enrollment on study.
Frequency of dose limiting toxicities (DLTs).The frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by type, severity (as defined by the NIH CTCAE, version 5.0), seriousness, duration, and relationship to study treatment. | 4 weeks
  For Cohort B, a Phase 1 run-in will be performed with the primary objective of evaluating the safety and tolerability of the combination of defactinib, avutometinib, and encorafenib in patients with BRAF V600E/K mutant melanoma with at least one untreated brain metastasis.
Response rate defined as Partial Response (PR) + Complete Response (CR) using Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria of all measurable target lesions present at the time of enrollment on trial. | 6 months
  For Cohort B, the primary objective will be to evaluate the preliminary response rate of the three drug combination of defactinib, avutometinib, and encorafenib in patients with BRAF V600E/K mutant melanoma. Measurable target lesions to be defined as all untreated and measurable (≥ 0.5 cm by 2 dimensional diameter measurements) present at the time of enrollment on study.

SECONDARY OUTCOMES:
Duration of response (DoR) | up to 5 years
  To assess the duration of response (DoR) of the study population. Duration of response is defined as the interval of time from the date of initial documented response (PR or better per Neuro-Oncology Brain Metastases (RANO-BM) criteria) to the time of progression from the best response, the start of a new therapy, or death
Disease control rate as defined by the proportion of subjects achieving a confirmed PR, CR, and SD as defined by Neuro-Oncology Brain Metastases (RANO-BM) criteria. | 6 months
  To assess the disease control rate in the study population.
Progression-free survival (PFS) as defined as the time from study drug initiation to the time documented disease progression (as assessed by Neuro-Oncology Brain Metastases (RANO-BM) criteria) or death from any cause. | up to 5 years
  To assess progression-free survival (PFS)
Time to development of new brain metastases as defined as the mean time from registration until development of new measurable (≥0.5 cm diameter) brain metastases not present on baseline MRI. | up to 5 years
  To assess the time to development of new brain metastases in the study population
Rate of new brain metastases defined as percent of study population that develop new measurable brain metastases between time of enrollment and time of documented progression (target or new lesions). | up to 5 years
  To assess the rate and frequency of development of new brain metastases of the study population. Frequency of new brain metastases defined as the number of new measurable brain metastases that develop in a particular patient between time of enrollment and time of documented progression (target or new lesions).
Overall survival (OS) defined as the time of study drug initiation until death from any cause | up to 5 years
  To assess overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Howard Colman, MD, PhD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No